CLINICAL TRIAL: NCT06666725
Title: Restaurant Menu Labeling: Added-sugar Labels and Labeling Thresholds
Brief Title: Effect of Added-sugar Menu Labels
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Davis (Other)
Responsible Party: Principal Investigator, Jennifer Falbe, Associate Professor, University of California, Davis
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Prevention
Other Study IDs: 1641776-8
Record Dates: First submitted 2024-10-17; First posted 2024-10-31 (Actual); Last update posted 2025-05-11 (Actual); Status verified 2025-05

CONDITIONS: Nutrition Knowledge; Dietary Behaviour

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (5):
- Control (No Intervention): Participant will order food and beverages from three menus. The menus will not contain any added sugar labels.
- Large, red, icon-only label, 50% daily value (Experimental): Participant will order food and beverages from three menus containing labels next to items that contain equal to or higher than half the daily value of added sugar (greater than or equal to 25 grams). The label will be on the right of the item, colored red, icon only design, and height that is 150% of size of the menu text height.
  Interventions: Other: Menu label
- Large, red, icon-only label, 100% daily value (Experimental): Participant will order food and beverages from three menus containing labels next to items that contain equal to or higher than the total daily value of added sugar (greater than or equal to 50 grams). The label will be on the right of the item, colored red, icon only design, and height that is 150% of size of the menu text height.
  Interventions: Other: Menu label
- Small, black, icon-plus-text label, 50% daily value (Experimental): Participant will order food and beverages from three menus containing labels next to items that contain equal to or higher than half the daily value of added sugar (greater than or equal to 25 grams). The label will be on the right of the item, colored black, icon plus text design, and height that is 100% of size of the menu text height.
  Interventions: Other: Menu label
- Small, black, icon-plus-text label, 100% daily value (Experimental): Participant will order food and beverages from three menus containing labels next to items that contain equal to or higher than the total daily value of added sugar (greater than or equal to 50 grams). The label will be on the right of the item, colored black, icon plus text design, and height that is 100% of size of the menu text height.
  Interventions: Other: Menu label

INTERVENTIONS:
Other: Menu label — Participants will select food items from three restaurant menus, displayed with labels as specified by their assigned group
  Arms: Large, red, icon-only label, 100% daily value; Large, red, icon-only label, 50% daily value; Small, black, icon-plus-text label, 100% daily value; Small, black, icon-plus-text label, 50% daily value

SUMMARY:
To compare two added-sugar menu label--(1) red, icon-only, 150% of the menu text height and (2) black, icon-plus-text, 100% of the menu text height--to a no-label control on grams of added sugar ordered using two different added-sugar labeling thresholds: (1) ≥50% of Daily Value for added sugar (equivalent to ≥25g) and (2) ≥100% of Daily Value for added sugar (equivalent to ≥50g)

DETAILED DESCRIPTION:
The main goal of this study is to compare two added-sugar menu labels--(1) red, icon-only, 150% of the menu text height and (2) black, icon-plus-text, 100% of the menu text height--to a no-label control on grams of added sugar ordered using two different added-sugar labeling thresholds: (1) ≥50% of Daily Value for added sugar (equivalent to ≥25g) and (2) ≥100% of Daily Value for added sugar (equivalent to ≥50g). This results in 5 conditions: (1) icon-only at 50% threshold, (2) icon-plus-text at 50% threshold, (3) icon-only at 100% threshold, (4) icon-plus-text at 100% threshold, and (5) no-label control.

The two primary outcomes are (1) grams of added sugar ordered averaged across a fast-food and full-service restaurant menus and (2) grams of added sugar ordered from a café menu. The secondary outcomes are (1) noticing a high added sugar nutrition label and (2) knowledge of items' added sugar content.

For continuous outcomes (e.g., grams of added sugar, knowledge), linear regression models regressing the outcome on an indicator for experimental condition will be used. If the outcomes are not normally distributed, alternative modeling approaches or data transformations will be explored. For dichotomous outcomes (e.g., noticing the added-sugar label), the probability ratio will be modeled using Poisson regression with a robust error variance, regressing the outcome on an indicator for experimental condition.

Exploration of effect modification of the labels on primary outcomes by type 2 diabetes status and sociodemographic variables important for health equity will be conducted using interaction terms and stratified models.

Exploratory process outcomes include (1) selection of at least one item that contains ≥50% of the Daily Value of added sugar and (2) selection of at least one item that contains ≥100% of Daily Value of added sugar. Other exploratory outcomes include the perception that the labels grabbed attention and support for an added sugars warning label policy. Additionally, differences in the primary outcomes between each of the 5 unique conditions will be examined. If there is evidence of interactions, the modeling approach will be modified.

ELIGIBILITY:
Inclusion Criteria:

* Equal or greater than 18 years of age
* English-speaking
* U.S. residents
* Have eaten restaurant food at least once in the last month
* Participants will reflect the U.S. Census Bureau's American Community Survey 5-year estimates for sex, race/ethnicity, educational attainment, and age

Exclusion Criteria:

* Failing the attention check question
* Completing the survey in less than 33% of the median completion time

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 11275 (Actual)
Dates: Start 2024-12-23 (Actual); Primary Completion 2025-02-13 (Actual); Study Completion 2025-02-13 (Actual)

PRIMARY OUTCOMES:
Grams of added sugar ordered averaged across fast-food and full-service menus | Within approximately 2 minutes of intervention exposure
  Continuous variable. Average grams of added sugar in foods and beverages selected, averaged across fast-food and full-service menus, analyzed using linear regression to examine differences between factor levels
Grams of added sugar ordered from a cafe menu | Within approximately 2 minutes of intervention exposure
  Continuous variable. Total grams of added sugar in menu items selected from a cafe menu, analyzed using linear regression to examine differences between factor levels

SECONDARY OUTCOMES:
Noticing and recall of added-sugar nutrient label - dichotomous variable "Correct" (Answered "Yes" to noticing, answered "Added sugars" to recall, and answered "high" for high low recall question) or "Incorrect" (otherwise) | Within approximately 10 minutes of intervention exposure
  Noticing a nutrition label - Measured with "Think back to the beginning of this survey when you imagined you were ordering dinner from restaurant menus. Did you notice any nutrition labels (other than the calories) next to any of the menu items?" Response options are "Yes", "No", and "Don't know".
  Recalling the label's meaning - [If answered "Yes"] Measured with "What did the nutrition label tell you about?" Response options are (displayed in survey in a random order) "Sodium", "Added sugars", "Trans fats", "Fiber", "Calcium", "Healthy items", "Unhealthy items", "Vegetarian", "Organic", "Gluten-free", "Sustainable", "None of these", "Not sure".
  High/low - [If answered "Added sugars"] "What did the label tell you about added sugars?" Response options are "High in added sugars", "Low in added sugars", "Something else", "I don't know".
  There is no formal name for this measure/scale.
Knowledge of menu items high in added sugar | Within approximately 10 minutes of intervention exposure
  Measured with "(While viewing menu excerpt) Click on the menu items that you think have equal to or more than half [or "equal to or more than the total", if assigned 100% threshold] the daily limit for added sugars." Continuous variable using the percent of 8 items correctly classified. Higher percentages of items correctly classified represent more knowledge.

OTHER OUTCOMES:
Selection of at least one item that has ≥50% of the Daily Value of added sugar | Within approximately 10 minutes of intervention exposure
  Dichotomous variable. "Yes" (ordered at least one that has ≥50% of the Daily Value of added sugar) or "No" (did not order any items high in added sugar), analyzed using Poisson regression.
Selection of at least one item that has ≥100% of Daily Value of added sugar | Within approximately 10 minutes of intervention exposure
  Dichotomous variable. "Yes" (ordered at least one that has ≥100% of Daily Value of added sugar) or "No" (did not order any items high in added sugar), analyzed using Poisson regression.

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Falbe, ScD, MPH, Principal Investigator — University of California, Davis
Locations (1):
- University of California, Davis, Davis, California, United States

IPD SHARING:
Plan to Share IPD: Yes
All variables used in the results of this study (experimental condition and individual level data on reactions to, perceptions of, and hypothetical behaviors in response to added-sugar menu label designs).
Time Frame: The IPD will be available no later than 6 months post-publication of all related research or 18 months from the end date of the award funding this work. The IPD will be available for approximately 5 years (depending constraints of the repository).
Access Criteria: Data will be deposited in an NIH-supported repository, access to which will be described on the principal investigator's website. A data sharing agreement will be required to ensure that the data will only be used for non-commercial research purposes.